CLINICAL TRIAL: NCT04601389
Title: An Open-label, Randomized, in Parallel Groups Comparative Study of Pharmacokinetics, Pharmacodynamics, Immunogenicity and Safety of Omalizumab (JSC "GENERIUM", Russia) and Xolair® ("Novartis Pharma AG", Switzerland) After Single-dose Subcutaneous Administration in Healthy Volunteers at 150 mg
Brief Title: Study of Pharmacokinetics, Pharmacodynamics and Safety Assessment of GNR-044 (JSC GENERIUM, Russia) and Xolair®
Acronym: NAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OMA-HVL-I; №88 eff.data 16 Feb 2017 (Registry Identifier: Ministry of Health of Russia approval number)
Record Dates: First submitted 2020-10-12; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Healthy Volunteers
Keywords: omalizumab; humanized monoclonal antibodies; total or free IgE; pharmacokinetics; pharmacodynamics; safety; bronchial asthma; health volunteers; equivalence; biosimilar; anti-allergic agents; anti-asthmatic agents; respiratory system agents; hypersensitivity; immune system diseases; urticaria
MeSH Terms: conditions — Asthma; Hypersensitivity; Immune System Diseases; Urticaria | interventions — Omalizumab

STUDY DESIGN:
Intervention Model Description: Interventional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GNR-044 (JSC "GENERIUM", the Russian Federation) (Experimental): 150 mg of omalizumab was subcutaneously injected once in the deltoid muscle area
  Interventions: Biological: Omalizumab (JSC "GENERIUM", the Russian Federation)
- Xolair® (Novartis Pharma AG, Switzerland) (Active Comparator): 150 mg of omalizumab was subcutaneously injected once in the deltoid muscle area
  Interventions: Biological: Xolair® (Novartis Pharma AG, Switzerland)

INTERVENTIONS:
Biological: Omalizumab (JSC "GENERIUM", the Russian Federation) — 150 mg of omalizumab was subcutaneously injected once in the deltoid muscle area
  Other Names: omalizumab; GNR-044
  Arms: GNR-044 (JSC "GENERIUM", the Russian Federation)
Biological: Xolair® (Novartis Pharma AG, Switzerland) — 150 mg of omalizumab was subcutaneously injected once in the deltoid muscle area
  Other Names: omalizumab
  Arms: Xolair® (Novartis Pharma AG, Switzerland)

SUMMARY:
An open-label, randomized, in parallel groups comparative study of pharmacokinetics, pharmacodynamics, immunogenicity and safety of GNR-044 (JSC "GENERIUM", Russian Federation) and Xolair® ("Novartis Pharma AG", Switzerland) after single subcutaneous administration in healthy volunteers at 150 mg

DETAILED DESCRIPTION:
There is an increasing incidence of bronchial asthma (BA) and other allergic diseases around the world. Bronchial asthma suffers from 4 to 10% of the world population, in Russian Federation, the incidence of BA across the adult population ranges from 2.2 to 5-7%, in the child population is about 10%.

Severe BA is associated not only with frequent hospitalizations and increased mortality but also with high treatment costs.

As to it, there is a hot button issue of developing new drugs for treating patients not to be achieved effectively with standard therapy. Considering the leading pathogenesis role of IgE-mediated allergy, the use of drugs to block IgE makes it possible to control the disease at the earliest allergic reaction phase of the development. It was shown that the IgE elimination from the mast cells and basophils surface reduced the severity of acute allergic reactions, reduced the allergen-induced late phase of the immune response and infiltration with inflammatory cells. These anti-IgE antibodies effects have been shown in various studies.

One of these drugs is оmalizumab (Xolair®). The drug has been approved in various countries across the world, including the United States and the European Union for the severe allergic BA and chronic idiopathic urticaria treatment. In the Russian Federation, omalizumab was registered in May 2007.

The drug GNR-044 (JSC "GENERIUM", Russian Federation) is biosimilar to the original drug Xolair®. This study is aimed to compare the safety and pharmacokinetics of the drug GNR-044 (JSC "GENERIUM", Russian Federation) and the drug Xolair® in order to register of the drug GNR-044 (JSC "GENERIUM", Russian Federation), a lyophilizate for subcutaneous administration, in the Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 50 (inclusive) at the time of the Informed Consent Form.
2. The diagnosis is "healthy" according to haematology and biochemical blood tests, urinalysis, results of physical examination, measurements of vital signs, results of electrocardiography.
3. Bodyweight from 40 to 90 kg inclusive.
4. Body mass index 18.5-30 kg / m2 inclusive.
5. Initial concentration of total IgE: ≥30 IU / ml and ≤300 IU / ml.
6. Comply with the rules of contraception by the study participants.

Exclusion Criteria:

1. Monoclonal antibodies administration within 1 year before taking omalizumab.
2. Hypersensitivity to any of the used study drug, to their components, history of an undesirable drug reaction.
3. Concurrent diseases and conditions with potential impact on the patient's safety, pharmacokinetics or pharmacodynamics.
4. The drug's use that affects pharmacokinetics or pharmacodynamics (injectable glucocorticosteroid drugs, allergen-specific immunotherapy, immunosuppressive drugs, vaccination within 30 days before signing informed consent and/or the need for vaccination during the study period).
5. Women of childbearing potential not using the contraception method(s), as well as women who are breastfeeding.
6. Patients with severe medical conditions that in the view of the investigator prohibits participation in the study.
7. Concurrent therapy with investigational agents.
8. A history of autoimmune disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the pharmacokinetic parameter - Tmax | 5-15 minutes before drug administration, in 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672, 984, 1344, 1680, 2016 hours after drug administration
  Tmax - Time to reach maximum concentration (day)
Assessment of the pharmacokinetic parameters - Cmax | 5-15 minutes before drug administration, in 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672, 984, 1344, 1680, 2016 hours after drug administration
  Cmax - Maximum concentration (μg / ml)
Assessment of the pharmacokinetic parameters - AUC0-∞ | 5-15 minutes before drug administration, in 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672, 984, 1344, 1680, 2016 hours after drug administration
  AUC0-∞ - Area under the concentration-time curve (mgday / ml) in the time interval from 0 to ∞
Assessment of the pharmacokinetic parameters - AUC0-2016 h | 5-15 minutes before drug administration, in 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672, 984, 1344, 1680, 2016 hours after drug administration
  AUC0-2016 h - Area under the concentration-time curve (mg day / ml) in the time interval from 0 to 2016 h
Assessment of the pharmacokinetic parameters - Kel | 5-15 minutes before drug administration, in 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672, 984, 1344, 1680, 2016 hours after drug administration
  Kel - Elimination constant (day - 1)
Assessment of the pharmacokinetic parameters - Vd/F | 5-15 minutes before drug administration, in 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672, 984, 1344, 1680, 2016 hours after drug administration
  Vd/F - Apparent volume of distribution (l)
Assessment of the pharmacokinetic parameters - CL/F | 5-15 minutes before drug administration, in 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672, 984, 1344, 1680, 2016 hours after drug administration
  CL/F - Apparent systemic clearance (ml / day)
Assessment of the pharmacokinetic parameters - T1/2 | 5-15 minutes before drug administration, in 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672, 984, 1344, 1680, 2016 hours after drug administration
  T1/2 - Half-life (day)
Assessment of the pharmacodynamics parameters - AUEC | 5-15 minutes before drug administration, in 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672, 984, 1344, 1680, 2016 hours after drug administration
  AUEC - (area under efficacy curve) the area under the curve "Relative difference in the free IgE concentration compared to the initial value - time"
Assessment of the pharmacodynamics parameters - Cmax | 5-15 minutes before drug administration, in 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672, 984, 1344, 1680, 2016 hours after drug administration
  Cmax - Maximum relative difference in free IgE concentration compared to baseline
Assessment of the pharmacodynamics parameters - relative difference estimation in free IgE concentration at each measurement point compared to baseline | 5-15 minutes before drug administration, in 6, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672, 984, 1344, 1680, 2016 hours after drug administration
  • relative difference estimation in free IgE concentration at each measurement point compared to baseline

SECONDARY OUTCOMES:
The frequency of antidrug antibodies formation | Before drug administration, on Day 15 ± 1 day, Day 42 ± 2 days and Day 85 ± 2 days after drug administration
  The frequency of antidrug antibodies formation
Antidrug antibody rate | Before drug administration, on Day 15 ± 1 day, Day 42 ± 2 days and Day 85 ± 2 days after drug administration
  Antidrug antibody rate
Neutralising antibodies rate | Before drug administration, on Day 15 ± 1 day, Day 42 ± 2 days and Day 85 ± 2 days after drug administration
  Neutralising antibodies rate
Body temperature measurement | Before drug administration, on Day 1-7, 11, 15, 22, 29, 42, 57, 71, 85 after drug administration
  A medical examination by an investigator to determine the state of a person's health, identify risk factors for AE and SAE: - body temperature measurement
Systolic blood pressure | Before drug administration, on Day 1-7, 11, 15, 22, 29, 42, 57, 71, 85 after drug administration
  A medical examination by an investigator to determine the state of a person's health, identify risk factors for AE and SAE: - systolic blood pressure
Diastolic blood pressure | Before drug administration, on Day 1-7, 11, 15, 22, 29, 42, 57, 71, 85 after drug administration
  A medical examination by an investigator to determine the state of a person's health, identify risk factors for AE and SAE: - diastolic blood pressure
Heart rate | Before drug administration, on Day 1-7, 11, 15, 22, 29, 42, 57, 71, 85 after drug administration
  A medical examination by an investigator to determine the state of a person's health, identify risk factors for AE and SAE: - heart rate
Respiratory rate | Before drug administration, on Day 1-7, 11, 15, 22, 29, 42, 57, 71, 85 after drug administration
  A medical examination by an investigator to determine the state of a person's health, identify risk factors for AE and SAE: - respiratory rate
Electrocardiogram (ECG) assessment of RR Interval | Before drug administration, on Day 29, 85 after drug administration
  A medical examination by an investigator to determine the state of a person's health, identify risk factors for AE and SAE - ECG RR Interval
Electrocardiogram (ECG) assessment of PQ Interval | Before drug administration, on Day 29, 85 after drug administration
  A medical examination by an investigator to determine the state of a person's health, identify risk factors for AE and SAE - ECG PQ Interval
Electrocardiogram (ECG) assessment of QRS Interval | Before drug administration, on Day 29, 85 after drug administration
  A medical examination by an investigator to determine the state of a person's health, identify risk factors for AE and SAE - ECG QRS Interval
Electrocardiogram (ECG) assessment of QT Interval | Before drug administration, on Day 29, 85 after drug administration
  A medical examination by an investigator to determine the state of a person's health, identify risk factors for AE and SAE - ECG QT Interval

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A Markova, MD, Study Chair — Head of the scientific department
Locations (2):
- Russia (2):
  - State budgetary institution of health care of the city of Moscow "City outpatients clinic No. 2 of the Department of Health of the city of Moscow", Moscow, RF
  - Federal State Budgetary Institution "State Scientific Center Institute of Immunology" by Federal Medical and Biological Agency of the Russian Federation, Moscow

IPD SHARING:
Plan to Share IPD: No
NAP

REFERENCES:
- See also: Clinical Trials Register — https://clinline.ru/reestr-klinicheskih-issledovanij/88-16.02.2017.html